CLINICAL TRIAL: NCT04629794
Title: The OsteoStrand Plus Deformity Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SeaSpine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SS-OS-1802
Record Dates: First submitted 2020-11-05; First posted 2020-11-16 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Spinal Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Demineralized Bone Matrix (Active Comparator): Prospective cohort subjects undergoing deformity correction surgery that receive Demineralized Bone Matrix (DBM).
  Interventions: Procedure: Posterolateral Lumbar Fusion with Demineralized Bone Fibers
- Bone Morphogenic Protein (Active Comparator): Retrospective cohort subjects that underwent deformity correction surgery and received Bone Morphogenic Protein (BMP).
  Interventions: Procedure: Posterolateral Lumbar Fusion with Bone Morphogenic Protein

INTERVENTIONS:
Procedure: Posterolateral Lumbar Fusion with Demineralized Bone Fibers — Posterolateral Lumbar Fusion with Demimeralized Bone Fibers
  Arms: Demineralized Bone Matrix
Procedure: Posterolateral Lumbar Fusion with Bone Morphogenic Protein — Posterolateral Lumbar Fusion with Bone Morphogenic Protein
  Arms: Bone Morphogenic Protein

SUMMARY:
A clinical study evaluating outcomes for patients with spinal deformity.

DETAILED DESCRIPTION:
A clinical study evaluating deformity patients treated with Demineralized Bone Matrix as compared to patients treated with Bone Morphogenetic Protein.

ELIGIBILITY:
Inclusion Criteria:

-≥18 years of age

* Indicated for deformity correction surgery
* Require spinal fusion at four or more levels
* Are willing to return for follow-up visits
* Willing to sign the Informed Consent Forms

Exclusion Criteria:

* Uncontrolled diabetes
* Morbid obesity
* history of alcohol or drug abuse
* Corticosteroid use
* Fever or leukocytosis
* Systemic infection
* Active malignancy
* Elevation of white blood cell count
* Osteoporosis
* Disease of bone metabolism
* Unsuitable or insufficient bone support
* Skeletal immaturity
* Prior fusion
* Use of steroids, immune suppressants, osteoporosis medications
* Use of internal bone stimulators
* Institutionalized or a prisoner
* Undergoing (Undergone) a worker's compensation case
* Pregnancy (includes women who are currently pregnant, lactating or wishing to become pregnant during the study duration)
* Participation in another research study involving another implant, product or drug that may affect the outcomes of this clinical study within the last 30 days, or planned during this clinical study
* Any other condition that the Investigator determines is unacceptable for enrollment into this clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of fusion for the demineralized bone matrix cohort vs bone morphogenic protein cohort | 12 Months
  Proportion of spinal levels in the demineralized bone matrix cohort vs bone morphogenic protein cohort achieving fusion.

SECONDARY OUTCOMES:
Clinical outcomes | 24 Months
  Oswestry Disability Index (ODI)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chang, MD, Principal Investigator — Sonoran Spine
Locations (1):
- Sonoran Spine, Tempe, Arizona, United States